CLINICAL TRIAL: NCT04155268
Title: Daily Assessments of Pain, Stress, and Sleep Following Flotation-REST: A Randomized Crossover Trial for Those With Chronic Pain
Brief Title: Flotation-REST for Chronic Pain, Stress, and Sleep
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to conduct the study due to Covid-19.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Steven Pratscher, Principal Investigator, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2017263
Record Dates: First submitted 2019-10-18; First posted 2019-11-07 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Healthy; Chronic Pain; Musculoskeletal Pain
Keywords: Healthy; Chronic Pain; Floatation-REST; Floating
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Floatation-REST (Experimental): Participants will float in a shallow pool of water with about 1000 pounds of epsom salt, in a light and sound attenuated device, for up to 60 minutes. Following the session, participants' ratings of the experience will be measured.
  Interventions: Behavioral: Flotation-REST
- Dark Room (Active Comparator): Participants will lay on an air mattress in a dark and quiet room, with reduced environmental stimulation, for up to 60 minutes. Following the session, participants' ratings of the experience will be measured.
  Interventions: Behavioral: Dark Room

INTERVENTIONS:
Behavioral: Flotation-REST — Floating in a specialized device (float pod or float cabin) used to attenuate sensory input.
  Arms: Floatation-REST
Behavioral: Dark Room — Participants will lay on an air mattress in a dark room with no cell phone and reduced sensory input.
  Arms: Dark Room

SUMMARY:
This randomized crossover trial aims to examine the effects of Flotation-REST (Reduced, Environmental, Stimulation, Technique/Therapy) compared to laying in a dark room (with reduced environmental stimulation) for those with chronic musculoskeletal pain. This design will allow for comparisons between the two interventions on daily diary assessments of pain, stress, and sleep, both between groups and within individuals.

DETAILED DESCRIPTION:
Chronic pain is a prevalent and significant health problem. Previous research shows that Flotation-REST may be an effective treatment for reducing pain but little is known about the short-term effects of a single session of Flotation-REST on the day-to-day variability of pain, stress, and sleep. Sleep, stress, and pain are all bidirectionally related to each other, and previous research shows that Flotation-REST may positively influence all three of these outcomes. Therefore, the primary aim of this study is to examine changes in pain, stress, and sleep following Flotation-REST. The secondary aim is to investigate whether various subjective experiences during the intervention are associated with changes in pain, stress, and sleep following the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Chronic musculoskeletal pain (e.g., back pain or upper or lower extremity pain, arthritis, fibromyalgia) on more days than not for the past 3 months
* Psychologically healthy
* Adults between the ages of 18-75 years.

Exclusion Criteria:

* Previous experience in a flotation-REST device.
* Diagnosed with neuropathic pain condition or endorsing more than 4 peripheral neuropathy symptoms.
* Diagnosed with any psychiatric condition (e.g., schizophrenia or bipolar disorder).
* Active suicidality with intent or plan.
* Currently taking SSRI medication.
* History of neurological conditions (e.g., epilepsy, stroke, severe traumatic brain injury, Parkinson's disease, Alzheimer's disease or other forms of dementia)
* Any skin conditions or open wounds that could cause pain when exposed to saltwater
* Inability to lay comfortably for 60 minutes
* Pregnant
* Started a new sleep or pain medication within the last 6 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-09 (Estimated); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Pain intensity | From baseline to follow-up, approximately 2 weeks
  Change in daily pain intensity where higher scores represent greater pain reduction using the Brief Pain Inventory
Pain Unpleasantness | From baseline to follow-up, approximately 2 weeks
  Change in daily pain unpleasantness where higher scores represent greater pain unpleasantness using the Brief Pain Inventory.
Stress | From baseline to follow-up, approximately 2 weeks
  Changes in perceived stress scale and daily diary assessments of stress where higher scores represent higher levels of stress.
Sleep | From baseline to follow-up, approximately 2 weeks
  Sleep Health Index and daily electronic dairies will be used to record sleep parameters. Higher sleep quality represents better sleep.

SECONDARY OUTCOMES:
Change in pain interference | From baseline to follow-up, approximately 2 weeks
  Change in daily pain interference where higher scores represent interference in daily activities from pain using the Brief Pain Inventory.
Change in muscle tension or tightness | Immediately before and after each intervention
  Average change in muscle tension from pre- to post-intervention where higher scores indicate greater muscle tension.
Change in self-actualization from baseline | Baseline, 1- week and 1-month after intervention
  Self-actualization Scale; 5-point Likert-type scale where the highest score indicates strongest self-actualization
Interoception | Immediately after each intervention
  Self-reported interoception assessed with the Multidimensional Interoceptive Awareness Scale after each intervention where higher scores indicate greater interoception during the session.
Insight | Immediately after each intervention
  Self-reported insights assessed with the Psychological Insight Questionnaire after each intervention where higher scores indicate more insight occurred during the session.
Emotional Breakthrough | Immediately after each intervention
  Self-reported emotional breakthrough assessed with the Emotional Breakthrough Inventory after each intervention where higher scores indicate more emotional breakthrough occurred during the session.
Mystical Experiences | Immediately after each intervention
  Self-reported mystical experiencesassessed with the Mystical Experiences Questionnaire after each intervention where higher scores indicate more mystical-type experiences occurred during the session.
Change in perceived stress | Baseline and 1-week after each intervention
  Perceived Stress Scale; assesses changes in perceived stress where higher scores indicate greater levels of stress
Change in Pain Catastrophizing | Baseline and 1-week after each intervention
  Pain Catastrophizing Scale; assesses changes in pain catastrophizing where higher scores indicate greater levels of pain catastrophizing
Change in Depression | Baseline and 1-week after each intervention
  Becks Depressive Inventory II; assesses changes in depression where higher scores indicate greater levels of depression
Persisting Effects | 1-week after each intervention
  Persisting Effects Questionnaire: scale of 0 - 5 where 5 is the strongest persisting effect

CONTACTS AND LOCATIONS:
Overall Officials: Steven Pratscher, Principal Investigator — University of Missouri-Columbia

IPD SHARING:
Plan to Share IPD: Undecided